CLINICAL TRIAL: NCT04533347
Title: A Double-blind Placebo-controlled Study to Assess the Efficacy and Safety of Oral Tafenoquine Versus Placebo in Patients With Mild to Moderate COVID-19 Disease
Brief Title: Tafenoquine in Patients With Mild to Moderate COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 60 Degrees Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQ 2020_06
Record Dates: First submitted 2020-08-28; First posted 2020-08-31 (Actual); Results first posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: COVID 19 Disease
Keywords: mild to moderate COVID 19 disease; SARS-CoV-2; infectious disease; severe acute respiratory syndrome coronavirus 2
MeSH Terms: conditions — Communicable Diseases | interventions — tafenoquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tafenoquine (Active Comparator): Tafenoquine two 100 mg oral tablets 1x/day on Days 1,2,3 and 10
  Interventions: Drug: Tafenoquine Oral Tablet
- Placebo (Placebo Comparator): Placebo two tablets 1x/day on Days 1,2,3 and 10
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tafenoquine Oral Tablet — Patients will be randomized and will receive and self-administer 200 mg Tafenoquine or matching placebo on Days 1, 2, 3, and 10.
  Other Names: ARAKODA™; KODATEF™
  Arms: Tafenoquine
Drug: Placebo — Patients will be randomized and will receive and self-administer 200 mg Tafenoquine or matching placebo on Days 1, 2, 3, and 10.
  Arms: Placebo

SUMMARY:
A clinical study to assess the efficacy and safety of oral tafenoquine compared to placebo in patients with mild to moderate COVID 19 disease.

DETAILED DESCRIPTION:
The TQ 2020_06 study is a double-blind placebo-controlled, Phase 2 clinical trial that plans to enroll approximately 275 patients with mild to moderate infection with COVID-19. Patients will undergo a brief screening period before being randomized to receive either self-administer 200 mg tafenoquine or matching placebo for 10 days. Following the treatment period, patients will have a follow up visit at study Day 28 (28 days after the first dose of study medication). The study's primary efficacy endpoint is proportion of patients with clinical recovery from COVID-19 symptoms on Day 14 in patients with mild to moderate COVID-19 disease compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥18 years of age;
* Laboratory confirmed infection with COVID-19 virus by an FDA-authorized SARS-Cov-2 RT-PCR;
* Able and willing to give written informed consent.
* Willing to keep an electronic diary from Study Day 1 to Study Day 13 (± 1 day) and Study Day 15 (± 1 day) to Study Day 28 (± 1 day)
* Willing to have daily phone or videoconferences with study team personnel from Study Day 1 to Day 13 (± 1 day) and Day 28
* At least one of the following clinical symptoms of COVID-19 infection within the 4 days prior to and inclusive of the day of screening:

  1. Respiratory rate ≥ 24/min
  2. New cough or shortness of breath that has presented within the last 4 days
  3. Fever - temperature 37.7°C [oral or skin surface]
* Must agree not to enroll in another study of an investigational agent prior to completion of Day 28 of the study.
* Able to take ARAKODA or KODATEF according to Prescribing Information
* Have been symptomatic no longer than 7 days when the first dose of study medication is administered.
* If female, agree to use an acceptable method of birth control from the time of consent through 56 days after the last dose of study drug.

Exclusion Criteria:

* Have one of the contraindications for ARAKODA or KODATEF in the prescribing information (section 16.1) including:

  1. G6PD deficiency
  2. Breastfeeding
  3. Psychotic disorder or current psychotic symptoms
  4. Known hypersensitivity reaction to TQ
* Evidence of severe or critical illness, defined by at least one of the following:

  1. Clinical signs indicative of severe systemic illness with COVID-19, such as respiratory rate ≥30 breaths per minute, heart rate ≥ 125 beats per minute, SpO2 ≤93% on room air
  2. Respiratory failure defined based on resource utilization requiring at least one of the following:

  i. Endotracheal intubation and mechanical ventilation, oxygen delivered by high flow nasal cannula (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates > 20 L/min with fraction of delivered oxygen ≥ 0.5), noninvasive positive pressure ventilation, extracorporeal membrane oxygenation (ECMO), or clinical diagnosis of respiratory failure (i.e., clinical need for one of the preceding therapies, but preceding therapies not able to be administered in setting of resource limitation) ii. Shock (defined by systolic blood pressure < 90 mmHg, or diastolic blood pressure <60 mmHg or requiring vasopressors) iii. Multi-organ dysfunction/failure
* Any other clinically significant acute illness unrelated to COVID-19 within seven days prior to first study drug administration
* Receipt of any experimental treatment for COVID-19 (off-label, compassionate use, or study-related) within the 30 days prior to the time of the screening evaluation
* Any excluded concomitant medication as described in the ARAKODA package insert [Section 16.1]. Receipt of a COVID-19 vaccine is not exclusionary.
* Any COVID-19 symptoms which, in the opinion of the investigator, is suggestive of possible requirement to hospitalize within 48 hours of enrollment
* Positive pregnancy test
* Have been symptomatic for more than seven days when the first dose would be administered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akila Chandrasekar, MD, Study Director — Peachtree BioResearch Solutions Inc.
Locations (10):
- United States (10):
  - Deluxe Health Center LLC, Miami, Florida
  - Hope Clinical Trials, Miami, Florida
  - F&T Medical Research, Inc., Miami, Florida
  - Kendall South Medical Center, Inc., Miami, Florida
  - Skyline Medical Center, Elkhorn, Nebraska
  - Burke Primary Care, Morgantown, North Carolina
  - AFC Urgent Care, Easley, South Carolina
  - Centex Studies, Brownsville, Texas
  - Care United, Forney, Texas
  - Clinical Trial Network, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geleris J, Sun Y, Platt J, Zucker J, Baldwin M, Hripcsak G, Labella A, Manson DK, Kubin C, Barr RG, Sobieszczyk ME, Schluger NW. Observational Study of Hydroxychloroquine in Hospitalized Patients with Covid-19. N Engl J Med. 2020 Jun 18;382(25):2411-2418. doi: 10.1056/NEJMoa2012410. Epub 2020 May 7. PMID 32379955
- [Background] Xiao F, Tang M, Zheng X, Liu Y, Li X, Shan H. Evidence for Gastrointestinal Infection of SARS-CoV-2. Gastroenterology. 2020 May;158(6):1831-1833.e3. doi: 10.1053/j.gastro.2020.02.055. Epub 2020 Mar 3. No abstract available. PMID 32142773
- [Background] Center for Disease Control. CDC Covid-19 data tracker. https://www.cdc.gov/covid-data-tracker/index.html#cases. Accessed March 7, 2020.
- [Result] Beigel JH, Tomashek KM, Dodd LE, Mehta AK, Zingman BS, Kalil AC, Hohmann E, Chu HY, Luetkemeyer A, Kline S, Lopez de Castilla D, Finberg RW, Dierberg K, Tapson V, Hsieh L, Patterson TF, Paredes R, Sweeney DA, Short WR, Touloumi G, Lye DC, Ohmagari N, Oh MD, Ruiz-Palacios GM, Benfield T, Fatkenheuer G, Kortepeter MG, Atmar RL, Creech CB, Lundgren J, Babiker AG, Pett S, Neaton JD, Burgess TH, Bonnett T, Green M, Makowski M, Osinusi A, Nayak S, Lane HC; ACTT-1 Study Group Members. Remdesivir for the Treatment of Covid-19 - Final Report. N Engl J Med. 2020 Nov 5;383(19):1813-1826. doi: 10.1056/NEJMoa2007764. Epub 2020 Oct 8. PMID 32445440
- [Result] Brueckner RP, Lasseter KC, Lin ET, Schuster BG. First-time-in-humans safety and pharmacokinetics of WR 238605, a new antimalarial. Am J Trop Med Hyg. 1998 May;58(5):645-9. doi: 10.4269/ajtmh.1998.58.645. PMID 9598455
- [Result] Crisafulli E, Clini EM. Measures of dyspnea in pulmonary rehabilitation. Multidiscip Respir Med. 2010 Jun 30;5(3):202-10. doi: 10.1186/2049-6958-5-3-202. PMID 22958431
- [Result] Dow GS, Luttick A, Fenner J, Wesche D, Yeo KR, Rayner C. Tafenoquine inhibits replication of SARS-Cov-2 at pharmacologically relevant concentrations in vitro. bioRxiv. January 2020:2020.07.12.199059. doi:10.1101/2020.07.12.199059
- [Result] Jia HP, Look DC, Shi L, Hickey M, Pewe L, Netland J, Farzan M, Wohlford-Lenane C, Perlman S, McCray PB Jr. ACE2 receptor expression and severe acute respiratory syndrome coronavirus infection depend on differentiation of human airway epithelia. J Virol. 2005 Dec;79(23):14614-21. doi: 10.1128/JVI.79.23.14614-14621.2005. PMID 16282461
- [Result] Skipper CP, Pastick KA, Engen NW, Bangdiwala AS, Abassi M, Lofgren SM, Williams DA, Okafor EC, Pullen MF, Nicol MR, Nascene AA, Hullsiek KH, Cheng MP, Luke D, Lother SA, MacKenzie LJ, Drobot G, Kelly LE, Schwartz IS, Zarychanski R, McDonald EG, Lee TC, Rajasingham R, Boulware DR. Hydroxychloroquine in Nonhospitalized Adults With Early COVID-19 : A Randomized Trial. Ann Intern Med. 2020 Oct 20;173(8):623-631. doi: 10.7326/M20-4207. Epub 2020 Jul 16. PMID 32673060
- [Result] Velavan TP, Meyer CG. The COVID-19 epidemic. Trop Med Int Health. 2020 Mar;25(3):278-280. doi: 10.1111/tmi.13383. Epub 2020 Feb 16. No abstract available. PMID 32052514
- [Result] Wang Y, Zhang D, Du G, Du R, Zhao J, Jin Y, Fu S, Gao L, Cheng Z, Lu Q, Hu Y, Luo G, Wang K, Lu Y, Li H, Wang S, Ruan S, Yang C, Mei C, Wang Y, Ding D, Wu F, Tang X, Ye X, Ye Y, Liu B, Yang J, Yin W, Wang A, Fan G, Zhou F, Liu Z, Gu X, Xu J, Shang L, Zhang Y, Cao L, Guo T, Wan Y, Qin H, Jiang Y, Jaki T, Hayden FG, Horby PW, Cao B, Wang C. Remdesivir in adults with severe COVID-19: a randomised, double-blind, placebo-controlled, multicentre trial. Lancet. 2020 May 16;395(10236):1569-1578. doi: 10.1016/S0140-6736(20)31022-9. Epub 2020 Apr 29. PMID 32423584
- [Result] Worldometer. Coronavirus Update (Live). https://www.worldometers.info/coronavirus/. Accessed March 7, 2020.
- [Result] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Mar;579(7798):270-273. doi: 10.1038/s41586-020-2012-7. Epub 2020 Feb 3. PMID 32015507

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tafenoquine | Placebo
Started | 45 | 41
Completed | 41 | 39
Not Completed | 4 | 2
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tafenoquine | Placebo | Total
Number analyzed (Participants) | 45 | 41 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (14.67) | 42.5 (14.76) | 42.6 (14.63)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years old | 20 | 17 | 37
  >= 40 years old | 25 | 24 | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 21 | 45
  Male | 21 | 20 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 30 | 65
  Not Hispanic or Latino | 10 | 11 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 43 | 41 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 45 | 41 | 86
Height [Mean (Standard Deviation); unit: centimeters] | 167.9 (10.60) | 167.0 (10.84) | 167.5 (10.67)
Height [Median (Full Range); unit: centimeters] | 167.6 [152 to 188] | 167.6 [140 to 188] | 167.6 [140 to 188]
Weight [Mean (Standard Deviation); unit: kilograms] | 82.6 (14.36) | 84.5 (22.68) | 83.5 (18.70)
Weight [Median (Full Range); unit: kilograms] | 81.0 [54 to 122] | 86.2 [48 to 145] | 82.3 [48 to 145]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Clinical Recovery of COVID-19 Symptoms on Day 14
Description: Clinical recovery from COVID-19 symptoms was defined as: temperature < or equal to 37.7 degrees Celsius (surface by infra-red or oral), respiratory rate < or equal to 24/minute on room air, shortness of breath is absent on a patient-report scale, and cough is mild or absent on a patient-reported scale.
Time Frame: Day 14 [± 1 day]
Population: Intention-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Tafenoquine | Placebo
Number analyzed (Participants) | 45 | 41
Participants
  Not Recovered | 8 | 10
  Recovered | 37 | 31
Statistical Analysis 1: Comparison: Tafenoquine vs Placebo; Assuming an 85% clinical recovery rate in the TQ group and a 70% clinical recovery rate in the placebo group, sample sizes of 125 per treatment group were expected to achieve 80% power with a two-sided alpha of 0.05; Test type: Superiority; p = 0.1879, Fisher Exact

2. Secondary Outcome: Increases the Proportion of Patients With Absence of Clinical Symptoms by Individual Symptom at Day 14
Description: Number and percentage of patients with COVID-19 clinical symptoms at Day 14 by individual symptoms (stuffy or runny nose, sore throat, shortness of breath, cough, low energy or tiredness, muscle or body aches, headache, chills or shivering, feeling hot or feverish, nausea, vomiting , diarrhea, sense of smell, and sense of taste)
Time Frame: Day 14 [± 1 day]
Measure: Count of Participants; unit: Participants
Arm/Group | Tafenoquine | Placebo
Number analyzed (Participants) | 45 | 41
Participants
  Stuffy or Runny Nose - None | 35 | 31
  Stuffy or Runny Nose - Mild | 6 | 6
  Stuffy or Runny Nose - Moderate | 1 | 2
  Stuffy or Runny Nose - Severe | 0 | 0
  Stuffy or Runny Nose - Not Done | 3 | 2
  Sore Throat - None | 39 | 37
  Sore Throat - Mild | 2 | 1
  Sore Throat - Moderate | 1 | 1
  Sore Throat - Severe | 0 | 0
  Sore Throat - Not Done | 3 | 2
  Shortness of Breath - None | 38 | 32
  Shortness of Breath - Mild | 4 | 6
  Shortness of Breath - Moderate | 0 | 1
  Shortness of Breath - Severe | 0 | 0
  Shortness of Breath - Not Done | 3 | 2
  Cough - None | 34 | 25
  Cough - Mild | 8 | 11
  Cough - Moderate | 0 | 3
  Cough - Severe | 0 | 0
  Cough - Not Done | 3 | 2
  Low Energy or Tiredness - None | 31 | 21
  Low Energy or Tiredness - Mild | 9 | 14
  Low Energy or Tiredness - Moderate | 1 | 3
  Low Energy or Tiredness - Severe | 1 | 1
  Low Energy or Tiredness - Not Done | 3 | 2
  Muscle or Body Aches - None | 37 | 32
  Muscle or Body Aches - Mild | 5 | 7
  Muscle or Body Aches - Moderate | 0 | 0
  Muscle or Body Aches - Severe | 0 | 0
  Muscle or Body Aches - Not Done | 3 | 2
  Headache - None | 34 | 33
  Headache - Mild | 6 | 5
  Headache - Moderate | 1 | 1
  Headache - Severe | 1 | 0
  Headache - Not Done | 3 | 2
  Chills or Shivering - None | 42 | 39
  Chills or Shivering - Mild | 0 | 0
  Chills or Shivering - Moderate | 0 | 0
  Chills or Shivering - Severe | 0 | 0
  Chills or Shivering - Not Done | 3 | 2
  Feeling Hot or Feverish - None | 41 | 39
  Feeling Hot or Feverish - Mild | 1 | 0
  Feeling Hot or Feverish - Moderate | 0 | 0
  Feeling Hot or Feverish - Severe | 0 | 0
  Feeling Hot or Feverish - Not Done | 3 | 2
  Nausea - None | 41 | 39
  Nausea - Mild | 1 | 0
  Nausea - Moderate | 0 | 0
  Nausea - Severe | 0 | 0
  Nausea - Not Done | 3 | 2
  How many times did you vomit in the last 24 hours? I did not vomit at all | 42 | 39
  How many times did you vomit in the last 24 hours? 1-2 times | 0 | 0
  How many times did you vomit in the last 24 hours? 3-4 times | 0 | 0
  How many times did you vomit in the last 24 hours? 5 or more times | 0 | 0
  How many times did you vomit in the last 24 hours? Not done | 3 | 2
  How many times did you have diarrhea in the last 24 hours? I did not have diarrhea at all | 39 | 37
  How many times did you have diarrhea in the last 24 hours? 1-2 times | 3 | 2
  How many times did you have diarrhea in the last 24 hours? 3-4 times | 0 | 0
  How many times did you have diarrhea in the last 24 hours? 5 or more times | 0 | 0
  How many times did you have diarrhea in the last 24 hours? Not done | 3 | 2
  Rate your sense of smell in the last 24 hours - My sense of smell is the same as usual | 19 | 17
  Rate your sense of smell in the last 24 hours - My sense of smell is less than usual | 18 | 19
  Rate your sense of smell in the last 24 hours - I have no sense of smell | 5 | 3
  Rate your sense of smell in the last 24 hours - Not done | 3 | 2
  Rate your sense of taste in the last 24 hours - My sense of taste is the same as usual | 20 | 15
  Rate your sense of taste in the last 24 hours - My sense of taste is less than usual | 19 | 21
  Rate your sense of taste in the last 24 hours - I have no sense of taste | 3 | 3
  Rate your sense of taste in the last 24 hours - Not done | 3 | 2

3. Secondary Outcome: Decreases the Hospitalization Rate Due to COVID-19 by Day 14
Description: Number and percentage of patients hospitalized due to COVID-19 symptoms (excluding non-COVID 19 causes including admittance for other upper respiratory infections and admittance only for administrative or observations purposes)
Time Frame: Day 14 [± 1 day]
Measure: Count of Participants; unit: Participants
Arm/Group | Tafenoquine | Placebo
Number analyzed (Participants) | 45 | 41
Participants | 1 | 2

4. Secondary Outcome: Decreases the Number of Medical Follow-up Visits by Day 14.
Description: Number and Percentage of Patients by Number of Medical Follow-up Visits (Doctor/ER Visit)
Time Frame: Day 14 [± 1 day]
Measure: Count of Participants; unit: Participants
Arm/Group | Tafenoquine | Placebo
Number analyzed (Participants) | 45 | 41
Participants
  Number of Doctor/ER Visits = 0 | 42 | 39
  Number of Doctor/ER Visits = 1 | 2 | 1
  Number of Doctor/ER Visits = 2 | 1 | 1
  Number of Doctor/ER Visits = 3 | 0 | 0
  Number of Doctor/ER Visits = 4 | 0 | 0
  Number of Doctor/ER Visits >=4 | 0 | 0

5. Other Pre Specified Outcome: Planned Interim Analysis and Data Monitoring
Description: Binding futility analysis of primary endpoint will be performed a minimum of 3 weeks after the earlier of [i] 100 pts. randomized or [ii] 6 months has elapsed since randomization of the first pt. in the study. Objective is to determine if tafenoquine increases the proportion of pts. with clinical recovery from COVID-19 symptoms on Day 14 in pts. with mild/moderate COVID-19 disease compared with placebo. Enrolment may be paused by sponsor prior to futility analysis if total number of pts. randomized reaches n=100 and re-initiated by sponsor after completion of futility analysis, if continuing study is determined to be non-futile. Unblinded interim analysis will be conducted by DMC statistician and results will be presented to DMC. If conditional power is less than the predetermined threshold, DMC will recommend terminating enrollment. Sponsor and study team will remain blinded, but will curtail enrollment based on recommendation of the DMC.
Time Frame: 100 patients randomized
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 28 days +/- 1 day
Arm/Group | Tafenoquine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/41
Serious Adverse Events (participants affected / at risk) | 1/45 | 2/41
Other Adverse Events (participants affected / at risk) | 8/45 | 4/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tafenoquine (N=45) | Placebo (N=41)
COVID-19 pneumonia (Infections and infestations) | 1 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tafenoquine (N=45) | Placebo (N=41)
Bronchitis (Infections and infestations) | 1 | 0
Transaminases increased (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Red blood cell count decreased (Investigations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT04533347/Prot_SAP_000.pdf